CLINICAL TRIAL: NCT01824238
Title: A 12-Week, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Assess the Efficacy and Safety of MK-0859 When Added to Ongoing Statin Therapy With or Without Other Lipid Modifying Therapies in Japanese Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study of the Safety and Efficacy of Anacetrapib (MK-0859) When Added to Ongoing Statin Therapy in Japanese Participants With Heterozygous Familial Hypercholesterolemia (MK-0859-050)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-050; 132234 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Heterozygous Familial Hypercholesterolemia (HeFH)
MeSH Terms: interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anacetrapib (Experimental): Participants will receive 100-mg anacetrapib tablet, orally, once-daily for 12 weeks.
  Interventions: Drug: Anacetrapib
- Placebo (Placebo Comparator): Participants will receive placebo tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo for anacetrapib

INTERVENTIONS:
Drug: Anacetrapib
  Other Names: MK-0859
  Arms: Anacetrapib
Drug: Placebo for anacetrapib
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of anacetrapib (MK-0859) on low-density lipoprotein-cholesterol (LDL-C) when compared to placebo in Japanese participants with heterozygous familial hypercholesterolemia when added to an existing statin lipid-modifying therapy.

ELIGIBILITY:
Inclusion Criteria:

* If female, cannot be of reproductive potential
* Diagnosed with heterozygous familial hypercholesterolemia
* Have been treated with an appropriate and

stable dose of statin± other lipid-lowering medication(s) for at least 6 weeks

Exclusion Criteria:

* Previously participated in a study with a cholesteryl ester transfer protein (CETP) inhibitor
* Homozygous familial hypercholesterolemia
* Severe chronic heart failure
* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery by-pass graft (CABG), unstable angina, or stroke within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in LDL-C (beta-quantification [BQ] method) | Baseline and Week 12
Percentage of Participants who Experience at Least One Adverse Event (AE) | 12 weeks

SECONDARY OUTCOMES:
Percent Change from Baseline in High-density Lipoprotein-cholesterol (HDL-C) | Baseline and Week 12
Percent Change from Baseline in Non-HDL-C | Baseline and Week 12
Percent Change from Baseline in Apolipoprotein A-I (Apo-A-I) | Baseline and Week 12
Percent Change from Baseline in Apolipoprotein B (Apo-B) | Baseline and Week 12
Percent Change from Baseline in Lipoprotein(a) (Lp[a]) | Baseline and Week 12

REFERENCES:
- [Result] Arai H, Teramoto T, Daida H, Ikewaki K, Maeda Y, Nakagomi M, Shirakawa M, Kakikawa T, Numaguchi H, Johnson-Levonas AO, Vaidya S, Blaustein RO. Efficacy and safety of the cholesteryl ester transfer protein inhibitor anacetrapib in Japanese patients with heterozygous familial hypercholesterolemia. Atherosclerosis. 2016 Jun;249:215-23. doi: 10.1016/j.atherosclerosis.2016.03.017. Epub 2016 Mar 25. PMID 27131642